CLINICAL TRIAL: NCT00204152
Title: Treatment for Chronic Depression With Behavioral Interventions
Brief Title: Treatment for Chronic Depression
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: PI left U of C
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 13166B
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Major Depressive Disorder
Keywords: Early onset depression; early adversity
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: (Condition 1) Behavioral Activation; (Condition 2) Behavioral Activation and Stress Innoculation

SUMMARY:
The purpose of this study is to test the clinical efficacy of two psychotherapies for early onset chronic major depression, including Behavioral Activation (Jacobson et al., 2001), and an integrated version of Behavioral Activation and Stress Innoculation Coping (BASIC) for short-term (16 weeks) of individual psychotherapy for adults with chronic major depression. The control condition is an individual workbook condition of Behavioral Activation. These psychotherapies focus on behavior activation, stress reduction and coping strategies to counter depressive symptoms.

DETAILED DESCRIPTION:
Early-onset unipolar major depression is linked with considerable morbidity and mortality (Birmaher et al., 1996). The goal of this project is to test the efficacy of Behavioral Activation (BA; Jacobson et al., 2001) and an integrated version of Behavioral Activation (BA + Stress Inoculation Coping; BASIC) for the short-term psychotherapy of adults with chronic major depression (onset before age 18) and a history of early life stress before age 18. Exposure to stress during the developmental years has been linked with early-onset depression (Rao et al., 1996), a propensity to generate stress during the life span (Hammen et al., 1998), and a greater psychological sensitivity to stress as an adult (Post et al., 1992). And while incidence of early life stress is high among depressed adults, there are no behavioral treatments designed to address the unique needs of these individuals. We aim to develop a new treatment for a specific group of depressed patients, namely individuals who report early onset of depression and early life stress. We include the critical elements of behavioral activation and stress reduction strategies to address the avoidance, stress sensitivities, and coping deficits often observed in this population.

The specific aims are: 1) to determine if the addition of stress reduction strategies (packaged in BASIC) enhance the effects of BA, as indexed by the rate early remission; 2) to investigate if exposure to BA and BASIC reduce risk of relapse within three months of treatment termination, as indexed by reduced rates of relapse by the 3-month follow-up; and, 3) to learn if effects of BA are mediated by changes in activity behaviors or the acquisition of compensatory behavioral skills, and likewise whether enduring effects of BASIC are mediated by changes in stress regulation or the acquisition of stress regulation skills. Our approach is to compare BA and BASIC to a self-guided bibliotherapy of BA (control condition) using a randomized clinical trial design to distinguish between conditions. We anticipate that this study will promote our understanding about the efficacy of BA and the discovery of mechanisms of treatment response. We expect this project to facilitate our understanding of the mechanisms that promote treatment gains and contribute to depressive relapse.

ELIGIBILITY:
Inclusion Criteria:

* depressed male and female subjects between ages 18 to 58 years.
* current and primary diagnosis of DSM-IV Major Depressive Disorder (e.g., no lifetime history of bipolar I or II disorder, current anxiety disorders, or current substance dependence disorder (American Psychiatric Association, 1994).
* should also have upon study entry a score of 14 or higher (moderate depression) on the Hamilton Rating Scale for Depression (HRSD; Hamilton, 1960) and a score of 20 or higher (moderate depression) on the Beck Depression Inventory II (BDI-II; Beck et al., 1996a).
* background of high childhood trauma (70-item Childhood Trauma Questionnaire with a Total Score of 9 or higher).
* reasonably fluent in English to complete the evaluation.

Exclusion Criteria:

* history of bipolar affective disorder,
* history of psychosis (including schizophrenia, schizophreniform disorder, schizoaffective disorder, delusional disorder, or psychotic organic brain syndrome)
* current non-psychotic Axis I disorder if it constitutes the predominant aspect of the clinical presentation and if it requires treatment other than that offered in the project (including anxiety disorders, somatoform disorders, dissociative disorders, or eating disorders, etc.),
* history of substance dependence in the past six months,
* antisocial, borderline, or schizotypal personality disorder,
* evidence of any medical disorder or condition that could cause depression or preclude the use of study treatments,
* current treatment with catecholaminergic antihypertensive medication, including reserpine, beta-blockers, clonidine, alphamethyldopa, etc. (diuretics, ACE inhibitors and calcium channel inhibitors will be allowed),
* clear indication of secondary gain (e.g., court ordered treatment or compensation issues),
* current suicide risk sufficient to preclude treatment on an outpatient basis (any patient scoring 3 or above on the suicide item on the HRSD or BDI must be cleared for study participation by the PI).

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2004-06; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
severity of depression, measured by Longitudinal Interval Follow-up Evaluation (LIFE; Keller et al., 1982; Keller et al., 1987), Beck Depression Inventory-II (BDI-II; Beck, Steer, & Brown, 1996a), and Hamilton Rating Scale for Depression.

SECONDARY OUTCOMES:
Cognitive functioning, social/behavioral functioning, and stress regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Jackie K Gollan, Ph.D., Principal Investigator — The University of Chicago, Department of Psychiatry
Locations (1):
- The University of Chicago, Department of Psychiatry, Chicago, Illinois, United States

REFERENCES:
- [Background] Jacobson NS, Dobson KS, Truax PA, Addis ME, Koerner K, Gollan JK, Gortner E, Prince SE. A component analysis of cognitive-behavioral treatment for depression. J Consult Clin Psychol. 1996 Apr;64(2):295-304. doi: 10.1037//0022-006x.64.2.295. PMID 8871414